CLINICAL TRIAL: NCT07014748
Title: SAFETY: Stabilization Points to Third Hospital Line Assessment oF the Impact of the usE of Infrascanner Model 2500 to Provide Decision Support for Diagnosis/Screening of Traumatic Brain InjurY in Ukraine
Acronym: SAFETY
Status: Recruiting | Type: Observational
Sponsor: InfraScan, Inc. (Industry)
Collaborators: USARMY USAMRMC (Unknown)
Responsible Party: Principal Investigator, Baruh Ben Dor, Principal Investigator, InfraScan, Inc.
Other Study IDs: 24-01-MPAI-179; 24-01-MPAI-179 (Other Grant/Funding Number: USARMY USAMRMC Combat Casualty Care)
Record Dates: First submitted 2025-05-22; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Hemorrhage
Keywords: TBI; ICH; Intracranial hematoma; Ukraine; Trauma; NIRS; Near Infrared
MeSH Terms: conditions — Brain Hemorrhage, Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Baseline Phase: Patients with suspected combat-related head trauma who are admitted to the participating hospitals will be eligible for enrollment in this trial. These patients will receive the current standard of care.
- Device Phase: Patients with suspected combat-related head trauma who are admitted to the participating hospitals will be eligible for enrollment in this trial. These patients will receive the current standard of care and the Infrascanner model 2500 will be added to the diagnosis and clinical decision.
  Interventions: Diagnostic Test: Handheld brain hematoma detector

INTERVENTIONS:
Diagnostic Test: Handheld brain hematoma detector — Near Infrared based handheld traumatic brain hematoma detector
  Other Names: Infrascanner Model 2500
  Groups: Device Phase

SUMMARY:
The Infrascanner model 2500 is a handheld, noninvasive device that is FDA-cleared to detect traumatic intracranial hematomas. FDA clearance K200203 was issued in 2020, K211617 added pediatric age group to the IFU in 2022, and K241389 approved higher laser power use to address dark skinned patients in 2024. This non randomized observational study aims to evaluate the utility of this device by evaluating its ability to provide decision support information to optimize care for patients with suspected traumatic intracranial hematomas. It is important to note that the intended use of the device is in accordance with its FDA approved indication. The intent is to generate actionable knowledge that along with standard clinical signs, facilitates the early detection of intracranial hemorrhage (ICH) in patients with suspected traumatic brain injury (TBI) in a combat setting. The ultimate goal is to modify and optimize international protocols for inexpensive, bedside, portable, and noninvasive detection of traumatic ICH in conflict zones across the globe.

This multicenter, prospective, observational, implementation science study will evaluate the field utility of the Infrascanner Model 2500 in an active combat setting using a pragmatic, sequential research design consisting of two phases-baseline phase and device phase. Using the current Ukrainian medical care system, patients with suspected TBIs will be monitored, and their outcomes will be tracked using standard-of-care practices (baseline phase). After the baseline data collection period is complete, an amendment to the protocol will be submitted to initiate the device phase. After training and upon approval, the Infrascanner device will be deployed to the facilities described above to provide health care providers with additional decision support, and the impact of its use will be compared to the baseline data. The outcome of interest is the time from admission at each enrollment study location to a definitive CT scan diagnosis of ICH. The investigators hypothesize that the use of the device will provide decision support to health care providers, decrease the time to traumatic ICH detection, thus enabling more expedient care.

This prospective study will include all patients with suspected combat-related head trauma identified by clinical signs of TBI, such as decreased GCS score, abnormal pupil exam, and/or asymmetrical motor exam, on admission to the clinical enrollment site (mobile hospital or regional clinical hospital) regardless of the presence of pharmacologic sedation. At the Vinnytsia hospital (Role 4), combat polytrauma preoperative patients will also be screened. Exclusion criteria include evidence of extensive scalp injury, including lacerations, avulsions, or abrasions that prevent proper placement of the Infrascanner device on a subject's head or prevent placement of the device in the specified locations.

During the baseline phase (Figure 1), 100 patients will be enrolled at stabilization points and the mobile/first-line hospital, 100 will be enrolled at the second-line hospital, and 100 will be enrolled at the third-line hospital. Thus, from a total of 300 subjects, baseline data on the time from admission at each enrollment study location to a definitive CT scan diagnosis of ICH and treatment and early outcomes will be collected.

Once the baseline phase is complete and the amendment for the device phase is approved, it will be initiated. During this device phase, the Infrascanner will be deployed to stabilization points and the three levels of care (mobile hospitals and regional clinical hospitals). Data collection will continue until 100 patients are enrolled in the device phase for the three levels of care. All data collection at the baseline and device phases will occur at the same locations, and the data elements will be identical, except for Infrascanner data collected during the device phase.

By comparing data from the baseline and device phase, the investigators will assess the utility of the device to provide decision support information to providers and potentially reduce time to definitive diagnosis by CT scan and thus treatment, as well as the association between Infrascanner use and early patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected combat-related head trauma identified by clinical signs of TBI on admission to the clinical enrollment site
* Clinical signs of TBI:

  * Decreased GCS score
  * Abnormal pupil exam
  * Asymmetrical motor exam
* The presence of pharmacologic sedation is not exclusion criteria.

Exclusion Criteria:

* Evidence of extensive scalp injury that prevent proper placement of the Infrascanner device on a subject's head or prevent placement of the device in the specified locations.
* Extensive scalp injury includes lacerations, avulsions, or abrasions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected combat-related head trauma
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Time from admission to definitive diagnosis | From admission at each enrollment study location to a definitive CT scan diagnosis of intracranial hemorrhage (ICH), which is up to 24 hours from admission.
  Evaluate the time from admission at each enrollment study location to a definitive CT scan diagnosis of intracranial hemorrhage (ICH).

SECONDARY OUTCOMES:
Final Glasgow Coma Scale at discharge or transfer | From admission to the hospital until 3 days from admission
  Evaluate the impact of Infrascanner data on early patient Glasgow Coma Scale changes
Number of Brain-related complications | From admission to the hospital until 3 days from admission
  Evaluate the impact of Infrascanner data on reduction of Brain-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Dmytro Dmytriiev, MD, PhD, MBA, Principal Investigator — Vinnytsia City Clinical Hospital named after M.I.Pirogov of Vinnitsya Regional Council
Locations (4):
- University of Alabama in Birmingham, Birmingham, Alabama, United States
- Ukraine (3):
  - Dnipropetrovsk Regional Clinical Hospital named after I.I. Mechnikov of Dnipropetrovsk Regional Council, Dnipro
  - Ukrainian Military, Kyiv
  - Vinnytsia City Clinical Hospital named after M.I.Pirogov of Vinnitsya Regional Council, Vinnytsia

IPD SHARING:
Plan to Share IPD: No
Most patients are members of the Ukrainian military and as a condition for the study a more severe data policy was accepted